CLINICAL TRIAL: NCT05894473
Title: Comparison of the Effects of Telerehabilitation-Based Motor and Cognitive Dual-Task Exercise in Patients With Parkinson's Disease - A Randomized Controlled Study
Brief Title: Effects of Telerehabilitation-Based Motor and Cognitive Dual-Task Exercise in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Ebru Akbuğa Koç, Assistant Professor, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor-Motor Dual Task Training Exercises (Active Comparator): Motor-Motor Dual Task Physical Exercises will be given to the participants
  Interventions: Other: Motor-Motor Dual Task Physical Exercises
- Cognitive-Motor Dual Task Training Exercises (Active Comparator): Cognitive-Motor Dual Task Physical Exercises will be given to the participants
  Interventions: Other: Motor-Motor Dual Task Physical Exercises
- Structured exercise program (Active Comparator): Physical exercise will be given to the participants
  Interventions: Other: Motor-Motor Dual Task Physical Exercises

INTERVENTIONS:
Other: Motor-Motor Dual Task Physical Exercises — Only physical exercise and motor dual tasks will be given

SUMMARY:
The ability to respond to multiple stimuli is impaired in Parkinson's patients. Traditional rehabilitation approaches focus only on balance and gait training, but individuals with Parkinson's disease need to perform multiple tasks in daily life.

DETAILED DESCRIPTION:
The dual-task (DT) methodology aims to perform two tasks simultaneously. There is no study in which motor and cognitive dual-task exercises are given together and followed up remotely in elderly individuals with PD.

Therefore, it was aimed to compare the effects of telerehabilitation method and motor and cognitive dual-task exercises on cognitive function, balance, walking, fall risk and quality of life in individuals with Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with idiopathic Parkinson's Disease

  * Getting at least 21 points from the Montreal Cognitive Assessment Scale test
  * Stability of drug therapy taken in the last 1 month
  * Being in the "ten" period of the patients
  * Being able to walk independently on flat ground (3 and above according to Functional Ambulation Classification)

Exclusion Criteria:

* • Serious hearing or vision problems

  * Having other neurological, cardiovascular or orthopedic disorders that may prevent walking
  * Any other neurological disorder (eg dementia, cerebrovascular disease)
  * Having an education level of less than 5 years
  * Patients with a pacemaker
  * Having vascular lower extremity pathologies
  * Not having internet access with a smart phone or computer

Ages: 40 Years to 87 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Parkinson's Disease Quality of Life Questionnaire | 8 weeks
  Parkinson's Disease Quality of Life Questionnaire
Montreal Cognitive Assessment Scale (MoCA) | 8 weeks
  Montreal Cognitive Assessment Scale (MoCA)
Berg Balance Scale (BBS) | 8 weeks
  Berg Balance Scale (BBS)
10 meter walking speed test | 8 weeks
  10 meter walking speed test
Timed Up And Go Test | 8 weeks
  Timed Up And Go Test
Fall Efficiency Scale - International | 8 weeks
  Fall Efficiency Scale - International
Five Times Sit to Stand Test | 8 weeks
  Five Times Sit to Stand Test

CONTACTS AND LOCATIONS:
Overall Officials: Yeditepe University, Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No